CLINICAL TRIAL: NCT04917627
Title: Randomized Controlled Trial Assessing Use of Vancomycin Powder in Craniotomy on Wound Infection Rates
Brief Title: To Assess Use of Vancomycin Powder in Craniotomy on Wound Infection Rates
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. sirajeddin belkhair, Head of department, neurosurgery, neuroscience institute, Hamad General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRC-01-18-220
Record Dates: First submitted 2021-05-21; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vancomycin group (intervention arm) (Active Comparator): We will use one vial of vancomycin that contains 1000 mg of the drug in powder form on the surgical site before closing the wound
  Interventions: Drug: Vancomycin
- control group (No Intervention): no vancomycin powder will be used

INTERVENTIONS:
Drug: Vancomycin — one vial of vancomycin (1000 mg ) powder form.
  Other Names: vancomax 1000mg powder form, KULLANMA TALİMATI
  Arms: vancomycin group (intervention arm)

SUMMARY:
Surgical site infection (SSI) after craniotomy is a major cause of morbidity and mortality besides its major health care cost. In each hospital, all measures are taken to decrease SSI. Despite current prophylactic measures, rates of SSIs have been reported in up to 5% of patients post craniotomy. Intrawound vancomycin powder has been studied extensively in spinal fusion surgeries and been found to reduce rates of surgical site infections (SSIs) significantly. Despite its success in spinal surgeries, topical vancomycin has not been extensively studied with respect to cranial neurosurgery.

The use of adjuvant vancomycin powder was associated with a significant reduction in the incidence of postoperative infection as well as infection-related medical costs. These findings suggest that the use of adjuvant vancomycin powder in high-risk patients undergoing spinal fusion is a cost-saving option for preventing postoperative infections, as it can lead to cost-savings of $438,165 per 100 spinal fusions performed.

The investigators believe that Topical vancomycin is a safe, effective, and cost-saving measure to prevent SSIs following craniotomy.

DETAILED DESCRIPTION:
its Prospective Randomized clinical trial. The investigator will do block randomization that is done by a biostatistician through SAS software . Patients will be divided in this Trial into two groups, first group (intervention arm) they will receive the drug (vancomycin). The second group (control arm) they will not receive the drug, otherwise both groups they will receive identical measure to decrease the postoperative SSI.

The investigator will use one vial of vancomycin that contains 1000 mg of the drug in the powder form.

The primary outcome variable will be SSI rate factored by cohort. Secondary outcome will be cost savings from vancomycin usage estimated from hospital costs associated with SSI in craniotomy patients, morbidity and mortality.

SSI found to be around 0.49% when vancomycin was used, while SSI in standard care found to be 5%, to get power of study 80% and level of significance 5%. Sample size will be 250 in each group using sample size calculator.

The statistical formula used in computation of required and adequate sample size in view of primary outcome i.e., SSI rate between the two groups:

The sample size was computed using the following statistical formula and sample size determination equation:

n = (Zα/2+Zβ)2 * (p1(1-p1)+p2(1-p2)) / (p1-p2)2

Where Zα/2 is the critical value of the Normal distribution at α/2 (e.g. for a confidence level of 95%, α is 0.05 and the critical value is 1.96), Zβ is the critical value of the Normal distribution at β (e.g. for a power of 80%, β is 0.2 and the critical value is 0.84) and p1 and p2 are the expected sample proportions of the two groups (SSI rate between the two groups i.e., vancomycin and control groups).

Before the study starts the investigator will do automated coded file with each code randomized to either arm (intervention arm and regular arm), then patient will be assigned to subsequent arm according to the code. CONSORT guidelines will be followed when reporting the results of the trail.

ELIGIBILITY:
Inclusion Criteria:

1. Any type of craniotomy whatever the cause.
2. Age more than 18 Years
3. Patient with no evidence of any source of infection

Exclusion Criteria:

1. Any evidence of infection.
2. Age less than 18 years
3. Previous and multiple craniotomies
4. Active infection
5. Craniectomy
6. wound laceration over the craniotomy site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
rate of wound infection | 24 months
  to assess the effectiveness of vancomycin in craniotomy on the surgical site infection rate as compared to controls.

SECONDARY OUTCOMES:
asses the rate wound complication | 24 months
  to assess the complications of intrawound vancomycin like seroma , long term benefit and cost effectiveness of vancomycin use on hospital stay and patient recovery, and to look for any other infection at 3 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: sirajeddin belkhair, Principal Investigator — Hamad General Hospital
Locations (1):
- Hamad General Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No